CLINICAL TRIAL: NCT02507986
Title: Mobile Phones in Cryptogenic Stroke Patients Bringing Single Lead ECGs to Detect Atrial Fibrillation
Acronym: MOBILE-AF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no personnel for recruitment
Sponsor: Leiden University (Other)
Collaborators: Medical Center Haaglanden (Other); Groene Hart Ziekenhuis (Other); Herning Hospital (Other); Alrijne Hospital (Other); Reinier de Graaf Groep (Other)
Responsible Party: Principal Investigator, Serge A. Trines, S.A.I.P. Trines, Senior Cardiologist, Leiden University Medical Center
Organization: Leiden University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MOBILE-AF
Record Dates: First submitted 2015-07-15; First posted 2015-07-24 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Atrial Fibrillation; Ischemic Stroke; Transient Ischemic Attack
MeSH Terms: conditions — Atrial Fibrillation; Ischemic Stroke; Ischemic Attack, Transient | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7-Day Holter monitor (Active Comparator): This arm will receive a 7-Day Holter monitor directly after randomization.
  Interventions: Device: 7-Day Holter monitor.
- Single lead ECG device (Experimental): This arm will be asked to take a single lead ECG two times per day and in case of complaints with a single lead ECG device.
  Interventions: Device: Single lead ECG device

INTERVENTIONS:
Device: Single lead ECG device — The single lead ECG device is a smartphone compatible handheld device that produces a single lead ECG after 30 seconds of measurement. It is non-invasive, electrically safe and easy to use.
  Arms: Single lead ECG device
Device: 7-Day Holter monitor. — The Holter is a conventional 7-Day Holter monitor.
  Arms: 7-Day Holter monitor

SUMMARY:
The main objective of this study is to compare the incidence of detected atrial fibrillation (AF) in cryptogenic stroke patients by a single lead ECG device with the incidence of detected AF by a 7-Day Holter ECG.

DETAILED DESCRIPTION:
Rationale: A standard work-up of stroke patients to identify a cause of stroke consists of Computed Tomography (CT), CT angiography of head and neck arteries, transthoracic echocardiography, 12-lead 10-seconds electrocardiogram (ECG), blood tests and 24-hour ECG monitoring. A stroke is called "cryptogenic" if no cause can be determined after standard work-up. Current detection of atrial fibrillation (AF) after stroke is 2.0%. Recent studies revealed that prolonged monitoring yields higher percentages of detected AF (12.0%). Devices used in these trials suffer from drawbacks. The investigators' hypothesis is that a new, smartphone compatible device, producing a single lead ECG (single lead ECG device), can be used for prolonged ECG monitoring in cryptogenic stroke patients.

Objective: The main objective of this study is to compare the incidence of detected AF in cryptogenic stroke patients by a single lead ECG device with the incidence of detected AF by a 7-Day Holter ECG.

Study design: A multicenter randomized trial. Study population: Cryptogenic stroke patients admitted to a hospital participating in the study. The calculated sample size is 200 (100 per arm).

Intervention: After inclusion, patients will be randomized to either a single lead ECG device or a 7-Day Holter Monitor.

Main study parameters/endpoints: The main endpoint will be the percentage of detected atrial fibrillation in both the single lead ECG device group and the 7-Day Holter group after one year.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Both devices are battery powered and electrically safe. Patients face a 2-3% risk that AF is detected false-positively; this might lead to incorrect oral anticoagulation (OAC) prescription. However, a potential benefit of the investigators' study is that if AF is detected and treated with OAC, this significantly reduces the chance of recurrent stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had an episode of symptomatic Transient ischemic attack (TIA) or episode of ischemic stroke.

  * Ischemic stroke is defined as an episode of transient or neurological dysfunction caused by focal brain or retinal ischemia with recent infarction on imaging
  * A TIA is defined as transient episode of neurologic dysfunction typically lasting less than one hour caused by focal brain or retinal ischemia without recent infarction on imaging.

Exclusion Criteria:

* Known etiology of TIA or ischemic stroke
* TIA or stroke caused by spinal ischemia
* TIA only presenting with non-localising symptoms
* Uncertainty about the diagnosis of TIA because of unclear clinical symptoms
* Myocardial infarction <6 months before stroke
* Coronary Artery Bypass Grafting <6 months before stroke
* Severe valvular heart disease
* Documented history of atrial fibrillation or atrial flutter
* Permanent indication for oral anticoagulation at enrolment
* Patient has permanent OAC contraindication
* Patient is included in another randomized trial
* Left ventricular aneurysm on echocardiography
* Thrombus on echocardiographyRenal dysfunction (creatinine clearance <30 mL/min/1.73m2)
* Patient has life expectancy of <1 year
* Patient is not willing to sign the informed consent form
* Patient is <18 years of age
* Patient is considered an incapacitated adult
* Patient is not in possession of a smartphone with Android Operating System (OS) or iOS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-07-29 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Percentage of detected atrial fibrillation | 1 year of follow-up

SECONDARY OUTCOMES:
Pro-Brain Natriuretic Peptide (Pro-BNP) levels in pg/mL | 24 hours after cryptogenic stroke
Percentages of atrial ectopy detected on 7-Day Holter monitor | 7 days after cryptogenic stroke
Left atrial diameter in cm/m2 | 24 hours after cryptogenic stroke
Number of participants with a recurrent stroke or TIA as defined in the trial | Within one year after cryptogenic stroke
Number of participants with a major bleeding | Within one year after cryptogenic stroke
Left atrial volume in mL/m2 | 24 hours after cryptogenic stroke

CONTACTS AND LOCATIONS:
Overall Officials: Serge Trines, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (7):
- Regionshospitalet Midtjylland, Herning, Denmark
- Netherlands (6):
  - Reinier de Graaf Hospital, Delft, South Holland
  - Groene Hart Ziekenhuis, Gouda, South Holland
  - Leiden University Medical Center, Leiden, South Holland
  - Alrijne Hospital, Leiderdorp, South Holland
  - Medisch Centrum Haaglanden, The Hague, South Holland
  - Bronovo ziekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Treskes RW, Gielen W, Wermer MJ, Grauss RW, van Alem AP, Dehnavi RA, Kirchhof CJ, van der Velde ET, Maan AC, Wolterbeek R, Overbeek OM, Schalij MJ, Trines SA. Mobile phones in cryptogenic strOke patients Bringing sIngle Lead ECGs for Atrial Fibrillation detection (MOBILE-AF): study protocol for a randomised controlled trial. Trials. 2017 Aug 29;18(1):402. doi: 10.1186/s13063-017-2131-0. PMID 28851409